CLINICAL TRIAL: NCT04516330
Title: Can MicroRNA's Predict Multicentricity in Breast Cancer?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Yeliz Emine Ersoy, Assoc. Prof., Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MCBC-MIR
Record Dates: First submitted 2013-12-10; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Multicentric Breast Cancer
Keywords: multicentric; breast; cancer
MeSH Terms: conditions — Neoplasms | interventions — MicroRNAs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- unifocal breast cancer (Active Comparator): patients having unifocal breast cancer
  Interventions: Genetic: miRNA
- multicentric breast cancer (Active Comparator): patients having multicentric breast cancer
  Interventions: Genetic: miRNA

INTERVENTIONS:
Genetic: miRNA — miRNA's expressed in breast cancer

SUMMARY:
The aim of this study is to determine if microRNA's have role in predicting multicentricity in breast cancer. If a specific microRNA will be found to be related with multicentricity, it will help us to make appropriate decisions on the treatment of patients with multicentric breast cancer.

DETAILED DESCRIPTION:
In the study that will be held at Bezmialem Vakif University Medical Faculty, General Surgery Department, 20 unifocal and 20 multifocal breast cancer patients will be included. Tissues will be taken from both tumoral and normal breast tissues and they will be saved in microRNA later solution under -80°C. Then, 84 microRNA's will be studied in these tissues to see if they express any of these microRNA's.

ELIGIBILITY:
Inclusion Criteria:

1. Having breast cancer
2. Having no other malignancy
3. Female patient

Exclusion Criteria:

1. Having other malignancy
2. Under 18 years old
3. Male patient

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-02; Primary Completion 2016-02 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
MicroRNA's in multicentric breast cancer | April 2014
  Evaluation of 84 microRNA's in patients with multicentric breast cancer

SECONDARY OUTCOMES:
Treatment plan according to the detected microRNA in patients with multicentric breast cancer | April 2014
  If a specific microRNA will be detected in patients with multicentric breast cancer, treatment plan will be individualized according to the detected microRNA

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)